CLINICAL TRIAL: NCT04745104
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Intravenous Administration of SHR-1707 in Healthy Young Adult and Elderly Subjects
Brief Title: A Trial of SHR-1707 in Healthy Young Adult and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1707-I-101-AUS
Record Dates: First submitted 2020-12-01; First posted 2021-02-09 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SHR-1707 Dose level 1 (Experimental): SHR-1707 or placebo is administered intravenous to young healthy subjects
  Interventions: Drug: SHR-1707; Drug: Placebo
- SHR-1707 Dose level 2 (Experimental): SHR-1707 or placebo is administered intravenous to young healthy subjects
  Interventions: Drug: SHR-1707; Drug: Placebo
- SHR-1707 Dose level 3 (Experimental): SHR-1707 or placebo is administered intravenous to young healthy subjects
  Interventions: Drug: SHR-1707; Drug: Placebo
- SHR-1707 Dose level 4 (Experimental): SHR-1707 or placebo is administered intravenous to young healthy subjects
  Interventions: Drug: SHR-1707; Drug: Placebo
- SHR-1707 Dose level 5 (Experimental): SHR-1707 or placebo is administered intravenous to young healthy subjects
  Interventions: Drug: SHR-1707; Drug: Placebo
- SHR-1707 Dose level 3 (Elderly subjects) (Experimental): SHR-1707 or placebo is administered intravenous to Elderly subjects
  Interventions: Drug: SHR-1707; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1707 — SHR-1707 will be administered through IV infusion
Drug: Placebo — Placebo will be administered through IV infusion

SUMMARY:
A randomized, double-blind, placebo-controlled, single dose escalation phase 1 study to access the Pharmacokinetics and Pharmacodynamics of Single Intravenous Administration of SHR-1707

DETAILED DESCRIPTION:
The study will consist of two parts: Subjects will be randomized to receive SHR-1707 as reflected by the guiding principle for the dose esclation/expansion phase. Each dose group includes a screening period, a baseline period, an observational period, and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial,
2. Male or female aged between 18 years and 45 years (inclusive) at the date of signed consent form in Part 1 and aged between 55 years and 80 years (inclusive) in Part 2
3. Total body weight of 45~100 kg (inclusive), with a body mass index (BMI) of 19~32 kg/m2 (inclusive) at screening and baseline
4. Subjects with good general health, no clinically significant abnormalities, or have underlying disease which is believed to have minimal impact on the study treatment in elderly subjects
5. WOCBP agree to take effective contraceptive methods

Exclusion Criteria:

1. Severe injuries or surgeries within 6 months before screening
2. ALT, or AST or total bilirubin level <1.5x upper limit of normal range (ULN) at screening or baseline visits
3. QTcF > 450msec (Male), QTcF > 470msec (Female) in 12-lead ECG test during screening and baseline
4. Known history or suspected of being allergic to the study drug.
5. Use of any medicine within 14 days (including any prescription, or over-the-counter medicine, herbal remedy or nutritional supplement, except for vitamins and acetaminophen with recommended dose [The dose of acetaminophen should be less than 2g/day, and no more than 3 days for continuous use]), or within 5 half-lives
6. Live (attenuated) vaccination within 1 month before screening
7. Blood donation or loss of more than 400 mL of blood within 3 months; or received blood transfusion within 3 months before screening.
8. History of alcohol abuse in the past 12 months of screening
9. History of illicit or prescription drug abuse or addiction within 12 months of screening
10. More than 5 cigarettes daily for 12 months before screening
11. Participation in clinical trials of other investigational drugs (include placebo) or medical devices within 3 months prior to screening
12. Researchers and relevant staff of the research center or other persons directly involved in the implementation of the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 12 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 12 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1707 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 12 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1707 administration
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 12 weeks)
  Time to Cmax of SHR-1707
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 12 weeks)
  Maximum observed concentration of SHR-1707
Pharmacokinetics-CL/F | Start of Treatment to end of study (approximately 12 weeks)
  Apparent clearance of SHR-1707
Pharmacokinetics-Vz/F | Start of Treatment to end of study (approximately 12 weeks)
  Apparent volume of distribution during terminal phase of SHR-1707
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 12 weeks)
  Terminal elimination half-life of SHR-1707
Pharmacokinetics MRT | Start of Treatment to end of study (approximately 12 weeks)
  Mean residence time of SHR-1707
Pharmacodynamics | Start of Treatment to end of study (approximately 12 weeks)
  Change from baseline of plasma biomarker concentrations
Anti-Drug antibody | Start of Treatment to end of study (approximately 12 weeks)
  The percentage of subjects with positive ADA titers over time for SHR-1707.

CONTACTS AND LOCATIONS:
Locations (1):
- Atridia Pty Limited, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Qiu H, Fan Y, Zhang Q, Qin H, Wu J, Zhang X, Liu Y, Zhou R, Zhang Q, Ye Z, Ma J, Xu Y, Feng S, Fei Y, Li N, Cui X, Dong F, Wang Q, Shen K, Shakib S, Williams J, Hu W. Safety, tolerability, pharmacokinetics and pharmacodynamics of a single intravenous dose of SHR-1707 in healthy adult subjects: two randomized, double-blind, single-ascending-dose, phase 1 studies. Alzheimers Res Ther. 2024 Oct 10;16(1):218. doi: 10.1186/s13195-024-01584-8. PMID 39390616